CLINICAL TRIAL: NCT00916487
Title: Efficacy of Fructose Metabolizing Enzymatic Product Fructosin(R) in Patients With Fructose Malabsorption
Brief Title: Efficacy of Fructose Metabolizing Enzymatic Product in Fructose Malabsorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciotec Diagnostic Technologies GmbH (Industry)
Collaborators: Austrian Research Promotion Agency (Other Government)
Responsible Party: Pongracz Christian, Sciotec Diagnostic Technologies GmbH
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fructo001; EUDRACT2008-005861-80
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Fructose Malabsorption
MeSH Terms: conditions — Fructose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm1 (Experimental): single arm of study in cross-over design
  Interventions: Dietary Supplement: Fructosin

INTERVENTIONS:
Dietary Supplement: Fructosin — Three capsules of Fructosin before one of the hydrogen breath tests.
  Other Names: Frutosin(R)

SUMMARY:
The purpose of this study is to determine whether the enzymatic product Frucosin(R) is able to degrade fructose in vivo in the small intestine of patients with known fructose malabsorption by measuring hydrogen in the expiratory air.

DETAILED DESCRIPTION:
Fructose malabsorption is a digestive disorder in which the uptake of fructose in the small intestine is deficient. This leads to an increase of the concentration of fructose in the large intestine after the intake of fructose-rich meals. The exzess fructose is then degraded by intestinal microbes into CO2, CH4, H2 and short chain fatty acids causing symptoms like bloating, diarrhea, flatulence or stomach pain.

The clinical diagnosis requires a hydrogen breath test after challenge with fructose. After an oral challenge with fructose the emerging hydrogen is measured in the expiratory air. A fructose malabsorption is diagnosed if the hydrogen in the expiratory air reaches 20ppm or more.

In the course of this study the participants will take 2 hydrogen breath tests. Before each of these tests the participants will take either the active treatment (Fructosin(R)) or a placebo. The active treatment should reduce the exhaled hydrogen indicating a reduced concentration of fructose in the large intestine after fructose metabolization by the verum.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed fructose malabsorption

Exclusion Criteria:

* Gravidity
* diabetes mellitus
* recent gastrointestinal surgery
* recent endoscopy
* recent antibiotics therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) of the exhaled breath hydrogen in ppm*min | 4 hours

SECONDARY OUTCOMES:
Symptoms during and after the hydrogen breath test (abdominal pain, flatulence, nausea and diarrhea/constipation) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Komericki, MD, Principal Investigator — Medical University of Graz; Christian Pongracz, MS, Study Director — Sciotec Diagnostic Technologies GmbH
Locations (1):
- Medical University of Graz, Graz, Styria, Austria